CLINICAL TRIAL: NCT05183802
Title: An Expanded Access Protocol for Setmelanotide for Treatment of Bardet-Biedl Syndrome (BBS)
Status: Approved for marketing | Type: Expanded Access
Sponsor: Rhythm Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: RM-493-036
Record Dates: First submitted 2021-11-08; First posted 2022-01-11 (Actual); Last update posted 2022-08-10 (Actual); Status verified 2022-08

CONDITIONS: Bardet-Biedl Syndrome (BBS); Obesity
MeSH Terms: conditions — Bardet-Biedl Syndrome; Obesity | interventions — setmelanotide

STUDY DESIGN:
Expanded Access Types: Treatment

INTERVENTIONS:
Drug: Setmelanotide, administered subcutaneously [SC], once daily. — Dosing based on age, and titrated from starting dose to target dose.

SUMMARY:
An open-label, single-arm, multicenter, Expanded Access Protocol [EAP] designed to provide treatment access to setmelanotide (3 mg, administered subcutaneously [SC], once daily) for eligible patients with BBS who have no alternative treatment options. All patients will continue to receive setmelanotide at the discretion of the Treating Physician and while they are deriving clinical benefit.

DETAILED DESCRIPTION:
This is an open-label, multicenter, EAP, designed to provide treatment access to setmelanotide for eligible patients who have BBS and who have no alternative treatment options.

Patients will undergo clinical and safety assessments before setmelanotide initiation, and then at 3 monthly intervals - or more frequently if clinically indicated - following initiation of setmelanotide and until treatment is completed or discontinued. All patients must have a 4 week (30 day) follow up safety evaluation after treatment is stopped.

The end of the program is defined as the last expected evaluation of the last patient or the date of reimbursement and commercialization of setmelanotide in these indications, whichever comes first.

ELIGIBILITY:
Patients who have not taken part in any previous setmelanotide clinical trial must fulfill all of the following study's eligibility criteria:

Inclusion Criteria:

1. Clinical diagnosis of BBS
2. Males and females aged ≥6 years
3. Obesity (≥30 kg/m2) for patients ≥18 years old or weight >97th percentile for age and sex on growth chart assessment for patients aged 6 to 17 years
4. Female participants of child-bearing potential must be confirmed as non-pregnant
5. Patients with significant neuropsychiatric disorders such as depression should be carefully evaluated regarding the benefit/risk ratio for the use of setmelanotide
6. Patients unable to enroll in another clinical trial with setmelanotide as determined by the treating physician

Exclusion Criteria:

1. Moderate to severe renal dysfunction defined as a glomerular filtration rate (GFR) <60 mL/min/1.73m2
2. History or close family history (parents or siblings) of skin cancer (excluding non-invasive basal or squamous cell lesion) melanoma, or patient history of ocular cutaneous albinism
3. Inability to comply with a daily injection regimen

Patients who have taken part in any previous setmelanotide clinical trial, have met all of the study's eligibility criteria, and have shown meaningful clinical benefit, defined as at least a 5% reduction in body weight for patients aged ≥18 years or a 5% reduction in BMI in patients aged <18 years from baseline through the end of the preceding study, will be eligible.

Min Age: 6 Years | Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Linda Shapiro, M.D., Ph.D., Study Chair — Chief Medical Officer, Rhythm Pharmaceuticals

REFERENCES:
- See also: Policy on Expanded Access to Investigational Drugs — https://www.rhythmtx.com/policy-on-expanded-access-to-investigational-drugs/